CLINICAL TRIAL: NCT03485391
Title: Peer Social Support During In Vivo Exposure for PTSD: A Program to Address Dropout From Prolonged Exposure
Brief Title: Peer Social Support During In Vivo Exposure for PTSD
Acronym: PEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Charleston Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00075914; W81XWH-18-1-0081 (Other Grant/Funding Number: U.S. Army Medical Research and Materiel Command)
Record Dates: First submitted 2018-03-07; First posted 2018-04-02 (Actual); Results first posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Stress Disorders, Post-Traumatic; Anxiety Disorders; Mental Disorder; Traumatic Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Mental Disorders; Wounds and Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PE+Exposure Workout Buddy (Experimental): Prolonged Exposure with assistance of Veteran who has successfully completed treatment to meet patients at exposure sites in the community to offer support during exposure.
  Interventions: Behavioral: Prolonged Exposure
- PE+Peer General Support (Active Comparator): Prolonged Exposure with assistance of Veteran who has successfully completed treatment to call and talk to patients once per week, informally meet at patient appointments, encourage session attendance and check in about progress.
  Interventions: Behavioral: Prolonged Exposure

INTERVENTIONS:
Behavioral: Prolonged Exposure — Practice guidelines have identified that trauma-focused psychotherapies have most evidence for treatment PTSD. Prolonged Exposure (PE) is one type of trauma-focused psychotherapy. PE teaches you to gradually approach trauma-related memories, feelings, and situations that you have been avoiding since your trauma. By confronting these challenges, you can decrease your PTSD symptoms. Treatment will last anywhere from 8-12 weeks for 75-90 minutes, once per week.

SUMMARY:
Veterans who have prematurely dropped out of exposure therapy for PTSD will be contacted and offered the opportunity to return to treatment, this time with the assistance of an in vivo exposure therapy 'workout buddy'. This peer will meet them at the in vivo exposure therapy location and offer support an encouragement while the patient remains in that location. As the PTSD treatment standards in Charleston and other VA sites across the country increasingly include telemedicine delivered care, both in person and telemedicine based exposure therapy recipients will be included. There will be no randomization; all participants will receive the peer support 'workout buddy' for exposure therapy assignments.

DETAILED DESCRIPTION:
Veterans (participants and peers) with PTSD will be recruited from the Charleston VA Medical Center catchment area. Participants will have been assigned to exposure therapy for PTSD and either started treatment, or dropped out before treatment; peers will have successfully completed exposure therapy for PTSD. Those eligible to participate will also include Veterans who are identified as "at-risk" of dropping out, Veterans who are uncomfortable completing in vivo exposure activities, and those who may have PTSD symptoms, but at the sub-threshold level. Participants will receive 8-12 weekly sessions of exposure therapy treatment with assistance of a PE Peer. Half of subjects will be randomized to the PE+Workout Buddy condition, where they will complete treatment with the assistance of a Veteran who will meet them at least once per week for in vivo exposure therapy assignments, for 3-4 weeks at the beginning of treatment. Half of subjects will be randomized to the PE+General Support condition, where they will complete treatment with the assistance of a Veteran who will call them via telephone once per week to encourage session attendance and ask about treatment progress, life stresses, etc. General support peers will also meeting Veterans 2-4 times per month to check in about treatment progress. All participants and peers will be consented. Participants will be assessed at baseline, post-treatment, and 3- & 6-month follow-up.

ELIGIBILITY:
Participant Inclusion Criteria:

1. Adult male or female over the age of 18 that has served, or is currently serving in the military.
2. Either diagnosis of PTSD as determined by a Clinician Administered PTSD Scale for DSM-5 (CAPS-5) clinical interview or CAPS-5 severity ≥ 25, and a PCL-5 score of ≥25.
3. Attempted PE treatment in the past, but did not complete treatment (defined as dropping out from treatment or refusal to engage in in vivo exposure assignments) OR identified as "at-risk" of dropping out of current exposure therapy treatment (defined as failure to complete 3 sessions of therapy within any 6 week period or verbally indicating that they are not comfortable with the exposure activities).

Participant Exclusion Criteria:

1. Active psychosis or dementia at screening.
2. Suicidal ideation with clear intent.
3. Concurrent enrollment in another clinical trial for PTSD or depression.

Peer Inclusion Criteria:

1. Adult male or female over the age of 18 that has served, or is currently serving, in the military.
2. Successful competition of exposure therapy treatment in the past and willingness to act as peer in the program.
3. PCL-5 score of 32 or lower.

Peer Exclusion Criteria:

1. Active psychosis or dementia at screening.
2. Suicidal ideation with clear intent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Muzzy, MRA, MLIS, Principal Investigator — Medical University of South Carolina; Ron Acierno, PhD, Principal Investigator — Ralph H. Johnson VA Medical Center
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Hernandez-Tejada MA, Muzzy W, Price M, Hamski S, Hart S, Foa E, Acierno R. Peer support during in vivo exposure homework to reverse attrition from prolonged exposure therapy for posttraumatic stress disorder (PTSD): description of a randomized controlled trial. Trials. 2020 Apr 28;21(1):366. doi: 10.1186/s13063-020-04302-5. PMID 32345329

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Specific inclusion criterion for patient-participants was a current diagnosis of PTSD as determined by the Clinician Administered PTSD Scale 5 (CAPS-5) or a CAPS-5 severity score ≥ 25, and a PTSD Checklist 5 (PCL-5) score of ≥ 25. Specific exclusion criteria were active psychosis or dementia, suicidal ideation with clear intent, and/or concurrent enrollment in another trial for PTSD or depression treatment.
Period: Overall Study
Arm/Group | PE+Exposure Workout Buddy | PE+Peer General Support
Started | 55 | 54
Completed | 38 | 34
Not Completed | 17 | 20

BASELINE CHARACTERISTICS:
Population: Participants were 109 Veterans aged 18 and over who were recruited from a southeastern Veterans Affairs Health Care System and its satellite Community Based Outpatient Clinics.
Groups:
- Total: Total of all reporting groups
Arm/Group | PE+Exposure Workout Buddy | PE+Peer General Support | Total
Number analyzed (Participants) | 55 | 54 | 109
Age, Continuous [Mean (Full Range); unit: years] | 43.6 [20 to 65] | 44.2 [22 to 74] | 43.9 [20 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 32 | 68
  Male | 19 | 22 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 7
  Not Hispanic or Latino | 49 | 52 | 101
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 31 | 22 | 53
  White | 18 | 29 | 47
  More than one race | 5 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 55 | 54 | 109

OUTCOME MEASURES:

1. Primary Outcome: Clinical Administrated PTSD Scale (CAPS)
Description: The Clinician Administered PTSD (Posttraumatic stress disorder) Scale (CAPS) is a 30-item structured interview that corresponds to the Diagnostic and Statistical Manual of Mental Disorders, 5th Version (DSM-V) criteria for PTSD. The CAPS can be used to make a current (past month) or lifetime diagnosis of PTSD or to assesses symptoms over the past week. CAPS-5 symptom cluster severity scores are calculated by summing the individual item severity scores for symptoms corresponding to a given DSM-5 cluster: Criterion B (items 1-5); Criterion C (items 6-7); Criterion D (items 8-14); and, Criterion E (items 15-20). A symptom cluster score may also be calculated for dissociation by summing items 19 and 20. Scores range from 0 to 80, with higher scores indicating worse outcomes.
Time Frame: 36 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PE+Exposure Workout Buddy | PE+Peer General Support
Number analyzed (Participants) | 55 | 54
score on a scale | 25.44 (11.966) | 24.44 (11.389)

2. Secondary Outcome: PTSD Checklist, 5th Version (PCL-5)
Description: The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. The PCL-5 has a variety of purposes, including, monitoring symptom change during and after treatment, screening individuals for PTSD, and making a provisional PTSD diagnosis. A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items (ranging from 0-4 per item). Higher scores indicate worse outcomes.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PE+Exposure Workout Buddy | PE+Peer General Support
Number analyzed (Participants) | 55 | 54
score on a scale | 32.1335 (18.77834) | 34.8677 (18.55918)

3. Secondary Outcome: PTSD Checklist, 5th Version (PCL-5)
Description: as for outcome 2
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PE+Exposure Workout Buddy | PE+Peer General Support
Number analyzed (Participants) | 55 | 54
score on a scale | 36.7449 (16.73793) | 34.8181 (16.53160)

4. Secondary Outcome: PTSD Checklist, 5th Version (PCL-5)
Description: as for outcome 2
Time Frame: 36 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PE+Exposure Workout Buddy | PE+Peer General Support
Number analyzed (Participants) | 55 | 54
score on a scale | 40.2105 (15.47735) | 37.1678 (17.18023)

5. Secondary Outcome: Patient Health Questionnaire (PHQ-9)
Description: The Patient Health Questionnaire -9 is widely used, well-validated measure of depression severity with high internal consistency (alpha .83 to .92; Cameron, Crawford, et al, 2008), and is correlated strongly with other depression measures. Its 9 items assess affective and somatic symptoms and correspond to diagnostic criteria for MDD. A total severity score (range - 0-27) can be obtained by summing the scores for each of the 9 items (ranging from 0-3 per item). Total scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively. Higher scores indicate worse outcomes.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PE+Exposure Workout Buddy | PE+Peer General Support
Number analyzed (Participants) | 55 | 54
score on a scale | 11.2105 (6.07833) | 11.5292 (5.83646)

6. Secondary Outcome: Patient Health Questionnaire (PHQ-9)
Description: as for outcome 5
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PE+Exposure Workout Buddy | PE+Peer General Support
Number analyzed (Participants) | 55 | 54
score on a scale | 12.0063 (5.36715) | 11.1333 (5.98522)

7. Secondary Outcome: Patient Health Questionnaire (PHQ-9)
Description: as for outcome 5
Time Frame: 36 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PE+Exposure Workout Buddy | PE+Peer General Support
Number analyzed (Participants) | 55 | 54
score on a scale | 12.5554 (5.17738) | 12.2859 (6.03785)

8. Secondary Outcome: Combat Exposure Scale (CES)
Description: The Combat Exposure Scale (CES) is a 7-item self-report measure that assesses wartime stressors experienced by combatants. Items are rated on a 5-point frequency (1 = "no" or "never" to 5 = "more than 50 times"), 5-point duration (1 = "never" to 5 = "more than 6 months"), 4-point frequency (1 = "no" to 4 = "more than 12 times") or 4-point degree of loss (1 = "no one" to 4 = "more than 50%") scale. Scores for each item are converted and then summed to obtain a total score. Total scores (of the converted items) range from 0 to 41, with lower scores indicating 'light' exposure and higher scores indicating 'heavy' exposure.
Time Frame: Baseline
Population: Over number of participants here vary slightly from the rest of the participant flow due to missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PE+Exposure Workout Buddy | PE+Peer General Support
Number analyzed (Participants) | 53 | 50
units on a scale | 4.1132 (5.97965) | 5.2400 (6.60723)

ADVERSE EVENTS:
Time Frame: Adverse event data collection started at baseline and progressed through treatment all the way to 6 month post treatment follow up. This time frame was 9 months.
Arm/Group | PE+Exposure Workout Buddy | PE+Peer General Support
All-Cause Mortality (participants affected / at risk) | 1/55 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/54
Other Adverse Events (participants affected / at risk) | 0/55 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT03485391/Prot_SAP_000.pdf